CLINICAL TRIAL: NCT07026513
Title: Observational Study on the Effectiveness of a First-line Therapy With Aminaphtone and Lidocaine Cream in Patients With Hemorrhoidal Disease: a Prospective Monocentric Cohort Study
Brief Title: ORal Aminaphtone and Combined LidocainE
Acronym: ORACLE
Status: Recruiting | Type: Observational
Sponsor: Treviso Regional Hospital (Network)
Responsible Party: Sponsor
Other Study IDs: ORACLE
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Hemorrhoid
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment - Aminaphtone + Lidocaine: Patients in this cohort receive a combination therapy with oral aminaphtone (Capillarema®: 1 tablet TID for 7 days, then BID for 3 weeks) and topical lidocaine cream (Octosedan®: at least twice daily or as needed) for 30 days. The goal is to assess symptom relief and tolerability of the combination as a first-line treatment for internal hemorrhoidal disease (Grade I-IV).
- Control - Standard Conservative Therapy: Patients in this cohort receive dietary and behavioral advice, including daily fiber intake (20-30 g/day) and hydration (≥1.5 L/day). They may also use topical Octosedan® and emollient creams as needed. This group represents guideline-based conservative management for symptomatic internal hemorrhoidal disease (Grade I-IV).

SUMMARY:
This observational study, called ORACLE (ORal Aminaphtone and Combined LidocainE), is being conducted at Treviso Regional Hospital (Italy) to evaluate the effectiveness of a first-line treatment for patients with internal hemorrhoidal disease (HD). The study focuses on a combination therapy using an oral drug, aminaphtone (Capillarema®), and a topical cream with lidocaine (Octosedan®), compared to standard conservative care.

Hemorrhoidal disease is a common condition that can cause bleeding, discomfort, itching, and swelling in the anal area. Many patients experience symptoms that affect their quality of life, even when using standard treatments like fiber supplements and emollient creams.

This study involves two groups of patients:

* One group will receive oral aminaphtone (Capillarema®) plus lidocaine cream (Octosedan®).
* The other group will receive standard advice on diet and hydration, along with optional use of lidocaine cream and emollients.

Patients will be followed for 30 days. The main goal is to measure how much the combination treatment improves hemorrhoidal symptoms compared to the standard treatment. This will be assessed using a score called HDSS (Hemorrhoidal Disease Symptom Score). The study will also evaluate quality of life using a specific questionnaire (SHS-HD) and assess how well patients tolerate the treatment.

About 50 adult patients will take part, divided into two consecutive groups of 25 each. The study does not involve random assignment or blinding. All participants will be informed about the study procedures and give written consent.

The results of this study may help doctors better understand the role of aminaphtone in managing hemorrhoidal disease and could improve future treatment recommendations.

DETAILED DESCRIPTION:
Detailed Description

The ORACLE study (ORal Aminaphtone and Combined LidocainE) is a prospective, monocentric, observational study designed to assess the real-world effectiveness and tolerability of a first-line therapy with aminaphtone (Capillarema®) and lidocaine cream (Octosedan®) in patients with symptomatic internal hemorrhoidal disease (HD). The study is conducted in a tertiary care hospital setting in Treviso, Italy.

Study Rationale

Hemorrhoidal disease affects up to 39% of the population, particularly between ages 45 and 65. Symptoms such as bleeding, anal pain, prolapse, and perianal swelling often result from vascular congestion and local inflammation. While conservative treatments including fiber intake and topical agents are frequently used, a substantial proportion of patients report persistent or recurrent symptoms.

Aminaphtone is a synthetic drug with well-documented endothelial-stabilizing and anti-inflammatory properties. It has been successfully used in the management of chronic venous insufficiency, diabetic microangiopathy, and Raynaud's phenomenon. Its mechanisms include modulation of adhesion molecules (e.g., VCAM-1, ICAM-1), pro-inflammatory cytokines (e.g., IL-6, VEGF, TGF-β), and vasoactive substances (e.g., endothelin-1). Given the similarities in vascular pathophysiology between hemorrhoidal disease and other chronic venous conditions, aminaphtone may offer therapeutic benefits in the hemorrhoidal setting.

Lidocaine, a well-established local anesthetic, is widely used for symptomatic relief in HD. The topical formulation (Octosedan®) included in this study is part of the standard conservative regimen in Italy.

Currently, there are no prospective studies evaluating the effectiveness of this combined regimen. The ORACLE study addresses this gap by comparing the combination therapy to standard conservative treatment in a real-world setting.

Study Design

This is a controlled, non-randomized, two-cohort study:

* Cohort A (Treatment group): Oral aminaphtone (Capillarema®) + topical lidocaine cream (Octosedan®)
* Cohort B (Control group): Standard conservative management (dietary advice, fiber, hydration, optional use of Octosedan® and emollient creams)

Participants will be enrolled in two consecutive time windows, with temporal allocation to either cohort. The duration of each participant's involvement is 30 days.

Inclusion Criteria

* Adults aged 18-85 years
* Symptomatic internal hemorrhoidal disease (Grade I-IV, Goligher classification)
* First outpatient consultation for current symptoms
* Written informed consent provided

Exclusion Criteria

* Concomitant proctologic conditions (e.g., fissures, fistulas, tumors)
* Inflammatory bowel disease
* HIV infection
* Previous surgical hemorrhoid treatment (unless >6 months prior and outpatient only)
* Current use of psychotropic, antibiotic, antifungal, immunomodulatory, or corticosteroid medications
* Known hypersensitivity to Capillarema® or Octosedan® components

Interventions

Treatment Group:

* Capillarema®: 1 tablet 3×/day for 7 days, then 2×/day for 3 weeks
* Octosedan®: ≥2 topical applications per day or as needed

Control Group:

* Dietary and behavioral advice
* Fiber intake: 20-30 g/day
* Hydration: ≥1.5 L/day
* Octosedan® and emollient creams as needed

Notably, the control arm does not include a placebo, as the conservative measures represent guideline-based first-line therapy per the Italian Society of Colorectal Surgery (SICCR).

Outcomes

Primary Endpoint:

* Change in HDSS (Hemorrhoidal Disease Symptom Score) from baseline (Day 0) to Day 30

Secondary Endpoints:

* Change in SHS-HD (Short Health Scale for Hemorrhoidal Disease)
* Local tolerability (burning, itching, pain) based on patient-reported symptoms and clinical assessment at Day 30

Sample Size

A total of 50 patients will be enrolled, 25 per cohort. This sample size assumes:

* A between-group difference in HDSS of 1.8 points
* Standard deviation (SD) of 1.7
* α = 0.05 and 90% power
* 10% expected dropout rate

Data Collection and Bias Mitigation

Data will be recorded using paper case report forms and transferred into a secure, anonymized database. To minimize bias, the follow-up visit will be performed by an investigator different from the one who conducted the baseline assessment.

Statistical Analysis

Primary analysis will follow both intention-to-treat and per-protocol principles. Statistical tests include:

* t-test or Mann-Whitney U test for continuous variables
* Chi-square or Fisher's exact test for categorical variables

Safety and Adverse Events

Adverse events (AEs) and serious adverse events (SAEs) will be recorded per ISO14155 guidelines, including severity and causal relationship with treatment.

Severity will be classified as:

* Mild: noticeable but tolerable symptoms
* Moderate: interferes with daily activities
* Severe: prevents normal activity

Causality terms:

* Certain
* Possible
* Not related

Ethical and Regulatory Considerations

The study will be conducted in accordance with the Declaration of Helsinki and Good Clinical Practice (GCP) guidelines (Ministerial Decree 15.07.97). Approval from the local Ethics Committee is required before study initiation. Written informed consent is mandatory.

Sponsorship and Conflict of Interest

This study is supported by an unrestricted grant from Laboratori Baldacci S.p.A., the manufacturer of Capillarema® and Octosedan®. The sponsor is not involved in study design, data analysis, or publication decisions.

Dissemination Plan

Findings from this study will be submitted for publication in peer-reviewed journals and presented at relevant scientific conferences. Trial results will also be updated on ClinicalTrials.gov in compliance with reporting requirements.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 85 years
* Diagnosis of symptomatic internal hemorrhoidal disease (Grade I-IV, Goligher classification)
* First outpatient consultation for current symptoms
* Written informed consent provided

Exclusion Criteria:

* Active proctologic conditions (e.g., anal fissures, fistulas, condylomas, neoplasms)
* Inflammatory bowel disease (IBD)
* Known HIV infection
* Previous surgical treatment for hemorrhoidal disease (except outpatient procedures performed >6 months prior)
* Current use of psychotropic, antibiotic, antifungal, immunomodulatory, or corticosteroid drugs
* Known hypersensitivity to Capillarema® or Octosedan® components

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-85 years) referred to the proctology clinic of Treviso Regional Hospital for a first evaluation of symptomatic internal hemorrhoids (Grades I-IV). Patients are consecutively enrolled in two non-randomized cohorts and represent a real-world outpatient population eligible for conservative treatment.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
HDSS | From baseline (Day 0) to Day 30
  Change in Hemorrhoidal Disease Symptom Score (HDSS) from baseline to Day 30. The HDSS is a validated tool that assesses the severity of five key symptoms of hemorrhoidal disease: pain, bleeding, itching, soiling, and prolapse. Scores range from 0 to 20.

CONTACTS AND LOCATIONS:
Locations (1):
- Regional Hospital Treviso, Treviso, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the monocentric nature of the study, the small sample size, and the absence of a data sharing infrastructure. Additionally, the informed consent obtained from participants does not include provisions for sharing anonymized data with external researchers. Any future data sharing would require a protocol amendment and additional ethics approval.